CLINICAL TRIAL: NCT06872476
Title: Influence of Bed Baths on Blood Gases and Vital Signs Given Under Heat to Children: Randomized Cross-Over Study
Brief Title: Bed Baths' Impact on Blood Gases and Vital Signs in Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nuh Naci Yazgan University (Other)
Collaborators: TC Erciyes University (Other)
Responsible Party: Principal Investigator, Dr. Zübeyde KORKMAZ, Assist. Prof Zübeyde KORKMAZ, Principal Investigator Pediatric Nursing, Department of Nursing, Faculty of Health Science., Nuh Naci Yazgan University
Allocation: Randomized | Model: Crossover | Purpose: Supportive Care
Other Study IDs: NuhNaciYazganU3
Record Dates: First submitted 2025-02-25; First posted 2025-03-12 (Actual); Last update posted 2025-03-12 (Actual); Status verified 2025-03

CONDITIONS: Vital; Blood Gases
Keywords: bed bath; blood gases; mechanical ventilator; pediatric intensive care; vital signs
MeSH Terms: interventions — Hot Temperature

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- bed bath (Experimental): This practice is a complementary and supportive care intervention.
  Interventions: Other: bed bath; Other: bed bath with heat
- bed bath with heat (Experimental): This practice is a complementary and supportive care intervention.In detail, this bed baths which were performed at under two heaters located 50-60 centimeters away from the bed of the children.
  Interventions: Other: bed bath; Other: bed bath with heat

INTERVENTIONS:
Other: bed bath
Other: bed bath with heat

SUMMARY:
Study Overview:

This randomized cross-over study investigated the effects of bed baths on the vital signs and blood gas values of children. The children received two bed baths: one under a heater and the other at room temperature. The order of the bed baths was randomized.

Methods:

The study involved children aged 1-36 months hospitalized in the Pediatric Intensive Care Unit (PICU). The bed baths were administered by a research nurse and assistant staff between 16:00 and 24:00 on weekends. The vital signs and capillary blood gas values (pH, PaO2, PaCO2, HCO3-) were measured three times: before, immediately after, and one hour after the bath. Data on heart rate, blood pressure, SpO2, and blood gas values were collected using specialized equipment.

Heating and Bathing Process:

For the heated bed bath, two heaters were positioned 50-60 cm above the child's bed, and the bath was conducted using soapy water at 37-40°C, followed by clear water.

Population:

The study was conducted in the PICU of a children's hospital, including children aged 1-36 months who were on mechanical ventilation, had normal body temperatures, and did not have chronic diseases. A total of 12 children participated over a period of two years.

Statistical Analysis:

Data were analyzed using IBM SPSS Statistics. Descriptive statistics such as percentages, averages, and standard deviations were used. The normality of the data was assessed, and repeated measurements were analyzed using ANOVA.

DETAILED DESCRIPTION:
Methods/Methodology This study was conducted in a randomized cross-over study. Study Design and Procedures In the study, children were given bed baths twice. One of the bed baths was done under heater and the other at room temperature. Which bed bath would be given first was determined by simple randomization (by lottery method). The bed baths of children participating in the study were given by a research nurse and an assistant staff. Children's bed baths are routinely given between 16:00 and 24:00 on weekends. Children who need a bed bath on weekdays are given a wiping bath by the caring nurse. The bed bath was performed in approximately at 21-240C room temperature in 20 to 25 minutes, with soapy water at 37-400C followed by clear water. The bed baths which were performed at under two heaters located 50-60 centimeters away from the bed of the children.

Measurements Applied at the Clinic The vital signs and capillary (right hand, middle finger) blood gas values were evaluated for a total of three times; five minutes before the bed bath, five minutes after the bed bath, and an hour after the bed bath.

1. Heart Rate Heart rates were measured using a PVM-2701 monitor (Nihon Kohden Corp., Tokyo, Japan).
2. Blood Pressure Blood pressures were measured manually over a period of one minute by a nursing team.
3. pH, PaO2, PaCO2 and HCO3- Measurements For all patients, pH, PaO2, PaCO2 and HCO3- measurements were recorded from capillary blood samples, using an ABL800 FLLEX blood gas analyzer (Radiometer Medical A/S, Brønshøj, Denmark).
4. SpO2 Measurements SpO2 was measured non-invasively using a PVM-2701 monitor (Nihon Kohden, Corp.). The saturation probe was applied to the patient's right palm. Daily measurements were recorded throughout each patient's stay in the Pediatric Intensive Care Unit (PICU).
5. Patient Warming To heat the environment during bathing, the heating devices (Patient Warming System, Nellcor) were fixed 50-60 centimeters upwards from the bed on two sides, both left and right Population and Samples The study was conducted in the PICU of the Children's Health Hospital affiliated with the Central Anatolian Public Hospitals Association. The intensive care unit where the study was conducted is an 8-bed 3rd degree PICU that cares for children between the ages of 1 month and 18 years. The data collection process took 2 years due to the long-term hospitalization of children in the unit and only children aged 1-36 months (Because of clinical nurses observed that the vital signs and blood gas values of children with mechanical ventilators for 1-36 months were affected after bedside bathing and that mechanical ventilator settings were changed) included in the study, and 12 children were reached in a two-year period. Children who are hospitalized for respiratory failures and in mechanical ventilators, not given Total Parenterally Nutrient, are normal body temperatures, are not suffering from any chronic diseases, and bathing would not cause problems was included.

Data Management and Statistical Analysis The data was evaluated in the IBM SPSS Statistics Standard Concurrent User V 25 (IBM Corp., Armonk, NY, USA) statistical package program. Number of units (n), percentage (%), average ± standard deviation (¯x±ss), median (M), and 25-75. percentile is given as descriptive statistics. Normal distribution of data regarding the numeric variables was evaluated with Q-Q plots and Shapiro-Wilk test for normality. Repeated measurements were variance analyzed (ANOVA).

ELIGIBILITY:
Inclusion Criteria:

* Children who are hospitalized for respiratory failures and in mechanical ventilators,
* having normal body temperatures

Exclusion Criteria:

* Total Parenterally Nutrition
* any chronic diseases
* any disease or condition which bathing would cause problems

Ages: 2 Months to 3 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 12 (Actual)
Dates: Start 2015-12-15 (Actual); Primary Completion 2017-12-30 (Actual); Study Completion 2018-03-15 (Actual)

PRIMARY OUTCOMES:
temperature measure | The bady temperature values were evaluated for a total of three times; five minutes before the bed bath, five minutes after the bed bath, and an hour after the bed bath. The values were measured three times in each bed bath, for a total of six times.
  Celcius
Pulse | The heart pulse values were evaluated for a total of three times; five minutes before the bed bath, five minutes after the bed bath, and an hour after the bed bath. The values were measured three times in each bed bath, for a total of six times.
  per minute
blood pressure | The blood pressure values were evaluated for a total of three times; five minutes before the bed bath, five minutes after the bed bath, and an hour after the bed bath.The values were measured three times in each bed bath, for a total of six times.
  mmHg
oxygen saturation | The oxygen saturation values were evaluated for a total of three times; five minutes before the bed bath, five minutes after the bed bath, and an hour after the bed bath. The values were measured three times in each bed bath, for a total of six times.
blood pH | The capillary blood pH values were evaluated for a total of three times; five minutes before the bed bath, five minutes after the bed bath, and an hour after the bed bath. The values were measured three times in each bed bath, for a total of six times.
  pH
PaO2 | The capillary blood PaO2 values were evaluated for total of three times; five minutes before the bed bath, five minutes after the bed bath, and an hour after the bed bath. The values were measured three times in each bed bath, for a total of six times.
PaCO2 | The capillary blood PaCO2 values were evaluated for a total of three times; five minutes before the bed bath, five minutes after the bed bath, and an hour after the bed bath.The values were measured three times in each bed bath, for total of six times.
HCO3- | The capillary blood HCO3- values were evaluated for a total of three times; five minutes before the bed bath, five minutes after the bed bath, and an hour after the bed bathThe values were measured three times in each bed bath, for total of six times.
  mEq/L

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kzl H, Sendir M. The Effects of Bed Bathing on Vital Signs and Oxygen Saturation in Children Who Are Connected to Mechanical Ventilation. Dimens Crit Care Nurs. 2018 Sep/Oct;37(5):272-278. doi: 10.1097/DCC.0000000000000312. PMID 30063523